CLINICAL TRIAL: NCT06327815
Title: Efficacy of FDC Regimen of Dapagliflozin/Metformin Compared to Co-administered Dual Therapy on Glycemic Control, Satisfaction and Adherence in Chinese Patients With T2DM: A 24-Week, Multicentre, Randomized, Parallel, Interventional, Non-inferiority, Open-label Study
Brief Title: Efficacy of FDC Regimen of Dapagliflozin/Metformin Compared to Co-administered Dual Therapy on Glycemic Control, Satisfaction and Adherence in Chinese Patients With T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690L00149
Record Dates: First submitted 2024-02-19; First posted 2024-03-25 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-administered Dual Therapy (Active Comparator): Dapagliflozin tablets and Metformin HCl extended-release tablets
  Interventions: Drug: Dapagliflozin tablets and Metformin HCl extended-release tablets
- FDC Regimen of Dapagliflozin/Metformin XR (Experimental): Xigduo (Dapagliflozin and Metformin hydrochloride extended-release) tablets
  Interventions: Drug: Xigduo (Dapagliflozin and Metformin hydrochloride extended-release) tablets

INTERVENTIONS:
Drug: Xigduo (Dapagliflozin and Metformin hydrochloride extended-release) tablets — 10 mg Dapagliflozin/1000 mg Metformin HCl extended-release
  Other Names: FDC Regimen of Dapagliflozin/Metformin XR
  Arms: FDC Regimen of Dapagliflozin/Metformin XR
Drug: Dapagliflozin tablets and Metformin HCl extended-release tablets — Dapagliflozin tablets: 10 mg Metformin HCl extended-release tablets: 1000 mg
  Other Names: Co-administered Dual Therapy
  Arms: Co-administered Dual Therapy

SUMMARY:
Study D1690L00149 is a 24-week, multicentre, randomized, parallel, interventional, non-inferiority, open-label study designed to compare the FDC Regimen of Dapagliflozin/Metformin XR with the Dapagliflozin co-administered with Metformin XR in glycemic lowering control, satisfaction and adherence in Chinese patients with T2DM.

DETAILED DESCRIPTION:
The past 30 years have witnessed significant increases in the prevalence of type 2 diabetes mellitus (T2DM) in China. China now is estimated 114 million people with diabetes, T2DM accounts for more than 90% of the overall population with diabetes in China. A large proportion of diabetes is undiagnosed in China: in the 2007-2008 national survey among adult population over 20 years, patient with newly diagnosed diabetes accounted for 60% of total diabetes population. In the Healthy China 2030 Plan, approved by the State Council and the Party's Central Committee, diabetes, along with cancer, hypertension, and cardiovascular diseases, are listed as the four major non-communicable diseases (NCDs) for which the goal is to "control the prevalence and reduce the probability of early death". Metformin hydrochloride is the primary biguanide medication currently used in China's medical practice. Sodium-glucose cotransporter 2 (SGLT2) inhibitors used to be considered as second-line treatment after Metformin in patients with T2DM. But according to the American Diabetes Association (ADA) 2023 Standards of Medical Care in Diabetes, SGLT2 inhibitors are now recommended to be started at the time of diagnosis as the first-line medications, for high-risk individuals with atherosclerotic cardiovascular disease (ASCVD), heart failure (HF) or chronic kidney disease (CKD). Compared with stepwise therapy, early combination therapy may provide earlier and greater reductions in HbA1c and thus achievement of glycemic target. In addition, SGLT2 inhibitors provide cardiorenal protection both in patients with and without T2DM, that goes beyond glycemic control, hence the recommendation by guidelines to implement SGLT2 inhibitors. But early combination therapy is not fully implemented into clinical practice in China. International and CDS guidelines recommends encourage using fixed-dose combination (FDC) to have better adherence, which is associated with lower HbA1c, lower cost and less need for acute care. But in practice, FDC is not popular in China because of many reasons. One of the main arguments is that physicians think FDC lacks flexibility. Compelling evidence has shown that the co-administration of Dapagliflozin and Metformin extended-release (XR) tablets is superior to either of the monotherapy efficacy (Dapagliflozin or Metformin XR). Xigduo XR combines those two anti-hyperglycemic medicinal products with different and complementary mechanisms of action to improve glycemic control in patients with T2DM. Bioequivalence was demonstrated between FDC regimen and coadministered Dapagliflozin and Metformin HCl XR tablets. This dosage of Dapagliflozin 10 mg/Metformin hydrochloride XR 1000 mg FDC (Xigduo XR) has no clinical evidence except that bioequivalence study in China, and there are no combination therapy data available either for Chinese people. (Metformin XR usual dose is 1500-2000mg/d). Moreover, there is no head-to-head study comparing Dapa/Met FDC and co-administration therapies to the extra benefits of FDC.

ELIGIBILITY:
Inclusion Criteria:

Age and Informed Consent

1. Patient must be 18 to 80 (years of age inclusive), at the time of signing the ICF(s).

   Type of Patient and Disease Characteristics
2. Newly diagnosed T2DM (WHO diagnostic criteria 1999) ≤ 1 year with medicine treatment naïve.
3. HbA1c 7.5%-10% at screening by local lab and HbA1c 7.5-10% at pre-randomization visit (by central laboratory).
4. BMI ≥19 and ≤40 kg/m2 at screening. Other Inclusion Criteria
5. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

Medical Conditions

1. Congestive heart failure NYHA classes III or IV or major cardiovascular events within 6 months before screening. (Significant cardiovascular history within the past 6 months prior to screening defined as: myocardial infarction, coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident.)
2. Patients with clinically apparent hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency. ALT or AST > 3x ULN, or serum TB >34.2 μmol/L (>2 mg/dL).
3. Patients with eGFR< 45 mL/min per 1.73 m².
4. Diagnosis or history of acute metabolic diabetic complications such as ketoacidosis or hyperglycemic hyperosmolar state, or diabetes insipidus within the past 6 months.
5. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
6. Participation in any other study that included drug treatment during the past 3 months before enrolment.

   Diagnostic Assessments
7. Patients with a known hypersensitivity to Dapa/Met or any of the excipients of the product.
8. Diagnosis or history of:

   1. Chronic pancreatitis within past 6 months or idiopathic acute pancreatitis within past 4 weeks.
   2. Gastrointestinal disease including gastroenterostomy, enterectomy, roemheld syndrome, severe hernia, intestinal obstruction, intestinal ulcer within past 6 months.
   3. Genetic galactose intolerance, lapp lactase deficiency and glucose-galactose malabsorption.
   4. Medullary thyroid carcinoma within past 5 years.
   5. Organ transplant or AIDS within the past 6 months.
   6. Alcohol abuse or illegal drug abuse within the past 12 months.
   7. Laser treatment for proliferative retinopathy within 6 months.
   8. Stress condition, such as surgery, serious trauma, etc., within past 6 months, or plan to undergo a surgery during study period.
   9. Chronic oxygen deficiency diseases, such as pulmonary emphysema, pulmonary heart disease within past 6 months.
   10. T1DM, diabetes resulting from pancreatic injury or secondary forms of diabetes, eg, acromegaly or Cushing's syndrome.

   Other Exclusions
9. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of study results.
10. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 24 weeks
  To demonstrate non-inferiority of Dapa/Met FDC regimen when compared with Dapa + Met co-administered with respect to the primary efficacy endpoint.

SECONDARY OUTCOMES:
Proportion of patients achieved HbA1c less than 7.0% from baseline to week 24. | 24 weeks
  To describe the changes from baseline at Week 24 in proportion of patients with HbA1c < 7%.
Absolute change in FPG from baseline to week 24. | 24 weeks
  To describe the changes from baseline at Week 24 in fasting plasma glucose (FPG).
Absolute change in PPG from baseline to week 24. | 24 weeks
  To describe the changes from baseline at Week 24 in postprandial glucose (PPG).
The difference in satisfaction scores between 2 groups measured with the Diabetes Treatment Satisfaction Questionnaire (DTSQ) at week 24. | Week 24
  To evaluate the difference in satisfaction of FDC versus co-administered dual therapy in Chinese patients with T2DM. The minimum value is 0, the maximum value is 36, higher scores mean a better outcome.
The difference in quality of life between 2 groups measured with Diabetes Quality of Life (DQOL) questionnaire at week 12 and week 24. | Week 12 and Week 24
  To evaluate the difference in quality of life of FDC versus co-administered dual therapy in Chinese patients with T2DM.
  DQOL-Satisfaction: the minimum value is 15, the maximum value is 75, higher scores mean a worse outcome.
  DQOL-Impact: the minimum value is 20, the maximum value is 100, higher scores mean a worse outcome.
  DQOL-Worry: the minimum value is 11, the maximum value is 55, higher scores mean a worse outcome.
To evaluate the difference in adherence of FDC versus co-administered dual therapy by Morisky Medication Adherence Scale-8 (MMAS-8) questionnaire in Chinese patients with T2DM. | Week 24
  To evaluate the difference in adherence of FDC versus co-administered dual therapy in Chinese patients with T2DM. The minimum value is 0, the maximum value is 8, higher scores mean a better outcome.

OTHER OUTCOMES:
AEs | 24 weeks
  An AE can therefore be any unfavourable and unintended sign (eg, an abnormal laboratory finding), symptom (for example nausea, chest pain), or disease temporally associated with the use of a medicinal product, whether it's considered related to the medicinal product.
SAE | 24 weeks
  An SAE is an AE occurring during any study phase (i.e., run-in, treatment, washout, follow up), that fulfils one or more of the following criteria:
  Results in death. Is immediately life-threatening. Requires in-patient hospitalization or prolongation of existing hospitalization.
  Results in persistent or significant disability or incapacity. Is a congenital anomaly or birth defect. Is an important medical event that may jeopardize the participant or may require medical treatment to prevent one of the outcomes listed above.
ADRs | 24 weeks
  An Adverse Drug Reaction (ADR) is an Adverse Event suspected to be causally related to the medicinal product.
Temperature | 24 weeks
  Armpit Temperature.
Systolic and diastolic BP | 24 weeks
  Blood pressure should be measured with a completely automated device in triplicate with at least 1-minute intervals between measurements after being comfortably at rest in a seated position(mmHg).
Pulse rate | 24 weeks
  Pulse rate should be measured with a completely automated device in triplicate with at least 1-minute intervals between measurements after being comfortably at rest in a seated position(times/min)
Respiratory rate | 24 weeks
  Respiratory rate per minute(times/min)
Weight | 24 weeks
  Weight in kilograms
Height | 24 weeks
  Height in meters
BMI | 24 weeks
  BMI in kg/m^2
Number of participants with abnormal ECG readings | 24 weeks
  The normality/abnormality of ECG tracings, as determined by the Investigator.
Proportion of TITR (Time in Tight Target Range) | Week 12
  The percentage of readings and time that a person spends with their blood glucose levels in a Tight target range (3.9-7.8mmol/L).
TIR (Time In Range) | Week 12
  The percentage of readings and time that a person spends with their blood glucose levels in a target range (3.9-10mmol/L).
TBR (Time Below Range) | Week 12
  The percentage of readings and time that a person spends with their blood glucose levels below target range.
TAR (Time Above Range) | Week 12
  The percentage of readings and time that a person spends with their blood glucose levels above target range.
MAGE (Mean Amplitude of Glycemic Excursion) | Week 12
  The mean of blood glucose values exceeding one SD from the 24-hour mean blood glucose and is used as an index of glycemic variability.
SDBG (Standard Deviation of Blood Glucose) | Week 12
  SDBG (Standard Deviation of Blood Glucose), reflects the amount of variation or dispersion of a series of glucose values.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, Principal Investigator — Beijing Chao Yang Hospital
Locations (31):
- China (31):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Chuxiong
  - Research Site, Dalian
  - Research Site, Dingzhou
  - Research Site, Fuyang
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hefei
  - Research Site, Jiangyin
  - Research Site, Jiyuan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Panjin
  - Research Site, Qingdao
  - Research Site, Quanzhou
  - Research Site, Rui’an
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Yibin
  - Research Site, Zhengzhou
  - Research Site, Zhuji

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Background] Boye KS, Curtis SE, Lage MJ, Garcia-Perez LE. Associations between adherence and outcomes among older, type 2 diabetes patients: evidence from a Medicare Supplemental database. Patient Prefer Adherence. 2016 Aug 16;10:1573-81. doi: 10.2147/PPA.S107543. eCollection 2016. PMID 27574406
- [Background] Han S, Iglay K, Davies MJ, Zhang Q, Radican L. Glycemic effectiveness and medication adherence with fixed-dose combination or coadministered dual therapy of antihyperglycemic regimens: a meta-analysis. Curr Med Res Opin. 2012 Jun;28(6):969-77. doi: 10.1185/03007995.2012.684045. Epub 2012 May 3. PMID 22494018
- See also: XIGDUO® XR PRESCRIBING INFORMATION FDA — http://www.accessdata.fda.gov/drugsatfda_docs/label/2022/205649s018lbl.pdf